CLINICAL TRIAL: NCT02194829
Title: A Phase I and Randomized Phase II Study of Nab-Paclitaxel/Gemcitabine With or Without AZD1775 for Treatment of Metastatic Adenocarcinoma of the Pancreas
Brief Title: Paclitaxel Albumin-Stabilized Nanoparticle Formulation and Gemcitabine Hydrochloride With or Without WEE1 Inhibitor AZD1775 in Treating Patients With Previously Untreated Pancreatic Cancer That Is Metastatic or Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01425; NCI-2014-01425 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2131 (Other: ECOG-ACRIN Cancer Research Group); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Results first posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Stage III Pancreatic Cancer AJCC v6 and v7; Stage IV Pancreatic Cancer AJCC v6 and v7; Unresectable Pancreatic Carcinoma
Keywords: Metastatic Pancreatic Adenocarcinoma; Nab-paclitaxel; Gemcitabine; AZD1775
MeSH Terms: interventions — adavosertib; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Patients also receive WEE1 inhibitor AZD1775 PO daily on days 1, 2, 8, 9, 15, and 16.
  Interventions: Drug: AZD1775; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Arm B (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor AZD1775 as in Arm A.
  Interventions: Drug: AZD1775; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: AZD1775 — Given PO
  Other Names: Adavosertib; MK-1775
Drug: Gemcitabine — Given IV
  Other Names: 2'-Deoxy-2'; 2'-difluorocytidine monohydrochloride; Gemzar
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI-007; paclitaxel protein-bound particles for injectable suspension

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of WEE1 inhibitor AZD1775 when given together with paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride and how well they work in treating patients with previously untreated pancreatic cancer that has spread to another place in the body or cannot be removed by surgery. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. WEE1 inhibitor AZD1775 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride are more effective with or without WEE1 inhibitor AZD1775 in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicity of combination therapy with nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation), gemcitabine (gemcitabine hydrochloride) and AZD1775 (WEE1 inhibitor MK-1775) in patients with treatment-naive metastatic adenocarcinoma of the pancreas or locally-advanced adenocarcinoma of the pancreas which is not surgically resectable. (Phase I) II. To determine the dose of AZD1775 to be used in combination with nab-paclitaxel and gemcitabine chemotherapy in the phase II portion of the trial. (Phase I) III. To determine the pharmacokinetics of AZD1775 in combination with nab-paclitaxel and gemcitabine. (Phase I) IV. To evaluate progression-free survival (PFS) associated with nab-paclitaxel/gemcitabine/placebo or nab-paclitaxel/gemcitabine/AZD1775 in patients with metastatic adenocarcinoma of the pancreas. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate overall survival (OS) associated with nab-paclitaxel/gemcitabine/placebo or nab-paclitaxel/gemcitabine/AZD1775 in patients with metastatic adenocarcinoma of the pancreas. (Phase II) II. To evaluate response rate (complete response [CR] + partial response [PR]) associated with nab-paclitaxel/gemcitabine/placebo or nab-paclitaxel/gemcitabine/AZD1775 in patients with metastatic adenocarcinoma of the pancreas. (Phase II) III. To evaluate disease control rate (CR + PR + stable disease [SD]) associated with nab-paclitaxel/gemcitabine/placebo or nab-paclitaxel/gemcitabine/AZD1775 in patients with metastatic adenocarcinoma of the pancreas. (Phase II)

TERTIARY OBJECTIVES:

I. To evaluate the ability of AZD1775 to inhibit Wee1 and increase deoxyribonucleic acid (DNA) damage and tumor cell death when combined with nab-paclitaxel/gemcitabine compared to nab-paclitaxel/gemcitabine/placebo. (Phase II) II. To evaluate if biomarker changes in tumor tissue associated with Wee1 inhibition may also be present in hair follicles. (Phase II) III. To evaluate the change in tumor fludeoxyglucose (FDG) uptake (maximum standardized uptake value [SUVmax]) between baseline FDG-positron emission tomography (PET) and week 4 FDG-PET as a predictor of response using Response Evaluation Criteria in Solid Tumors (RECIST) as the reference standard for response. (Phase II) IV. To evaluate the change in tumor FDG uptake (SUVmax) between baseline FDG-PET and week 4 FDG-PET as a predictor of progression-free survival. (Phase II) V. To compare the change in tumor FDG uptake (SUVmax) between baseline FDG-PET and week 4 FDG-PET between the patients from treatment arms C and D. (Phase II) VI. To evaluate if an early increase in tumor fluorothymidine (FLT) uptake (FLT-flare) is observed within 24 hours after initiation of treatment with nab-paclitaxel/gemcitabine/placebo. (Phase II) VII. To evaluate if an early (within 24 hours [h]) increase in tumor FLT uptake (FLT-flare) is abrogated after initiation of treatment with nab-paclitaxel/gemcitabine/AZD1775. (Phase II) VIII. To compare the change in tumor FLT uptake (SUVmax) from baseline to 24 hours after initiation of treatment between the patients from treatment arms C and D. (Phase II)

OUTLINE: This is a phase I, dose escalation study of WEE1 inhibitor AZD1775 followed by a randomized phase II study. Patients in phase I are assigned to arm A or B and patients in phase II are randomized to arm C or D.

ARM A (PHASE I, DOSE LEVEL 1): Patients receive paclitaxel albumin-stabilized nanoparticle formulation intravenously (IV) over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Patients also receive WEE1 inhibitor AZD1775 orally (PO) daily on days 1, 2, 8, 9, 15, and 16.

ARM B (PHASE I, DOSE LEVEL -2): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor AZD1775 as in Arm A.

ARMS C - G (PHASE I, DOSE LEVEL -1 to DOSE LEVEL 4): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor AZD1775 as in Arm A at various dose levels. These arms did not enroll any patients.

ARM H (PHASE II, Control): Patients receive paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride as in Arm A. The study did not move forward to the phase II part.

ARM I (PHASE II, WEE1 INHIBITOR AZD1775): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor AZD1775 as in Arm A. The study did not move forward to the phase II part.

In all arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria (Phase I):

* Patients must have histologically or cytologically confirmed metastatic or unresectable locally advanced adenocarcinoma of the pancreas. Prior therapy with a non-gemcitabine based regimen is permitted.
* Previous neo-adjuvant or adjuvant treatment is allowed provided that it was given >= 6 months prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have a life expectancy of >= 12 weeks
* Patients may have had prior radiotherapy for metastatic disease as long as it was > 4 weeks prior to registration and the patient has recovered from adverse events associated with the radiotherapy
* Patients must be able to swallow capsules whole
* Patients must be able to tolerate computed tomography (CT), magnetic resonance imaging (MRI) or PET imaging including contrast agents
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal and barrier method of birth control; two barrier methods of birth control; abstinence) for the duration of study treatment and for 3 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; should a man impregnate or suspect that he has impregnated a woman while participating in this study, he should inform his treating physician immediately
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal (ULN) or =< 5 X ULN if the patient has liver metastases
* Creatinine =< 1.5 mg/dL or creatinine clearance (Cockcroft-Gault) >= 60 mL/min for patients with creatinine levels above institutional upper limit of normal (ULN)

Exclusion Criteria (Phase I):

* Receiving any other investigational agents concurrently
* Have received any other investigational agents =< 4 weeks prior to registration
* Pre-existing > grade 1 motor or sensory neuropathy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nab-paclitaxel, gemcitabine or AZD1775
* Major surgical procedures <=28 days of beginning study treatment or minor surgical procedures <=7 days
* Taking current medications or substances that are inhibitors of CYP3A4, inhibitors or substrates of P-glycoprotein or inhibitors of breast cancer resistance protein (BCRP)
* Uncontrolled serious medical illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* Patients with known human immunodeficiency virus (HIV) and cluster of differentiation (CD)4 count is =< 200 cell/mm^3 or receiving antiretroviral therapy due to potential unfavorable interaction of the agents with the study treatment
* Previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, breast cancer in situ, or superficial bladder cancer (noninvasive papillary carcinoma or carcinoma in situ)
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years
* Pregnant or breast-feeding

  * Females of childbearing potential must have a blood test or urine study within 5 days prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* At least18 years of age

Inclusion Criteria (Phase II):

* Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas
* Patients must have measurable disease outside of the primary tumor (pancreas) by RECIST 1.1 criteria; baseline measurements and evaluations of all sites of disease must be obtained =< 4 weeks prior to randomization
* Previous neo-adjuvant or adjuvant treatment is allowed provided that there was no evidence of recurrent disease for at least 6 months after completion of neo-adjuvant/adjuvant treatment
* Patients may have had prior radiotherapy for metastatic disease as long as it was > 4 weeks prior to randomization and the patient has recovered from adverse events associated with the radiotherapy
* ECOG performance status of 0 or 1
* Life expectancy of >= 12 weeks
* Patients must be able to swallow capsules whole
* Patients with biliary stents are allowed
* Patients must be able to tolerate CT, MRI or PET imaging including contrast agents
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal and barrier method of birth control; two barrier methods of birth control; abstinence) for the duration of study treatment and for 3 months after the last dose of study treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; should a man impregnate or suspect that he has impregnated a woman while participating in this study, he should inform his treating physician immediately
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN)
* AST (SGOT)/ALT (SGPT) =< 3 X institutional upper limit of normal (ULN) or =< 5 X ULN if the patient has liver metastases
* Creatinine =< 1.5 mg/dL or creatinine clearance (Cockcroft-Gault) >= 60 mL/min for patients with creatinine levels above institutional upper limit of normal (ULN)
* For participation in the imaging research studies, patients must meet the additional following criteria:

  * The patient is participating in the trial at an institutional which has agreed to perform the imaging research studies, completed the American College of Radiation Imaging Network (ACRIN) defined scanner qualification procedures and received ACRIN approval
  * The patient has consented in writing to participate in one of the imaging research studies
  * The patient meets the criteria required for the imaging study in which the site is participating:

    * NOTE: Eligibility for participating in either imaging sub-study will depend on the availability of the imaging sub-study at a particular institution
  * For participation in the FDG-PET sub-study:

    * Patients must have an evaluable lesion of > 20 mm in size on standard practice imaging study as assessed by site (either primary pancreas mass or metastasis)
  * For participation in the FLT-PET sub-study:

    * Patients must be able to lie still for a 1.5 hour PET scan.
    * Patients must have an evaluable lesion in the pancreas > 20 mm in size on standard practice imaging study as assessed by site (lesion must be likely primary adenocarcinoma of the pancreas that is not primarily fibrotic or mucinous in nature)

Phase II Exclusion Criteria:

* Prior systemic therapy for metastatic disease
* Locally advanced disease
* Major surgical procedures <=28 days of beginning study treatment or minor surgical procedures <=7 days
* Any of the following cardiac diseases at registration or within the last 6 months as defined by New York Heart Association (NYHA) ≥ Class 2:

  * Unstable angina pectoris
  * Congestive heart failure
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication
  * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible.)
* Taking current medications or substances that are inhibitors of CYP3A4, inhibitors or substrates of P-glycoprotein or inhibitors of breast cancer resistance protein (BCRP)
* Prior Wee1 inhibitors or AZD1775
* Prior gemcitabine or nab-paclitaxel in a metastatic setting
* Corrected QT interval QTc > 470 msec (as calculated per institutional standards) at study entry or congenital long QT syndrome).
* Receiving any other investigational agents concurrently or have received any other investigational agents =< 4 weeks prior to randomization
* Pre-existing > grade 1 motor or sensory neuropathy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nab-paclitaxel, gemcitabine or AZD1775
* Uncontrolled serious medical illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements
* Previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, breast cancer in situ, or superficial bladder cancer (noninvasive papillary carcinoma or carcinoma in situ)
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years
* Pregnant or breast-feeding

  * Females of childbearing potential must have a blood test or urine study within 5 days prior to randomization to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* For participation in the FDG-PET sub-study:

  * Poorly controlled diabetes (defined as fasting glucose level >= 200 mg/dL) despite efforts to improve glucose control by fasting duration and adjustment of medications
  * Weigh more than the maximum weight limit for the PET table
* For participation in the FLT-PET sub-study:

  * History of allergic reaction attributable to compounds of similar chemical or biologic composition to 18F-fluorothymidine
  * Weigh more than the maximum weight limit for the PET table

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Eads, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 patients were enrolled between August 19, 2014 and November 1, 2016.
Groups:
- Arm A (Phase I - Initial Dose Level): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Patients also receive WEE1 inhibitor AZD1775 PO daily on days 1, 2, 8, 9, 15, and 16.
- Arm B ((Phase I - Dose Level -2): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor AZD1775 as in Arm A.
Period: Overall Study
Arm/Group | Arm A (Phase I - Initial Dose Level) | Arm B ((Phase I - Dose Level -2)
Started | 2 | 6
Received Protocol Therapy | 2 | 5
Completed | 0 | 0
Not Completed | 2 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Death | 0 | 1
Not completed — Disease progression | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Never started protocol therapy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only patients who started protocol therapy were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Phase I - Initial Dose Level) | Arm B ((Phase I - Dose Level -2) | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Continuous [Median (Full Range); unit: years] | 70.5 [68 to 73] | 73 [39 to 76] | 73 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT)
Description: A dose-limiting toxicity (DLT) was defined by the occurrence of any of the toxicities listed in section 5.1.5 of the protocol that are possibly, probably, or definitely related to study drug(s) within the first cycle (4 weeks = 28 days).
Time Frame: Assessed at 28 days
Population: Only patients who received protocol therapy were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B (Phase I - Dose Level -2): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor AZD1775 as in Arm A.
Arm/Group | Arm A (Phase I - Initial Dose Level) | Arm B (Phase I - Dose Level -2)
Number analyzed (Participants) | 2 | 5
Participants | 2 | 2

2. Primary Outcome: To Determine the Pharmacokinetics of AZD1775 in Combination With Nab-paclitaxel and Gemcitabine
Description: Plasma was to be collected on Cycle 1 Day 1 and Cycle 1 Day 16 for the pharmacokinetics analysis.
Time Frame: Assessed at Day 1 and Day 16
Population: Insufficient plasma samples were collected on this study so no pharmacokinetics analysis of AZD1775 in combination with nab-paclitaxel and gemcitabine was performed. Data were not collected. Consequently, no pharmacokinetics results of AZD1775 would be reported here.
Arm/Group | Arm A (Phase I - Initial Dose Level) | Arm B (Phase I - Dose Level -2)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Progression-free Survival
Time Frame: Assessed every 3 months for 2 years
Population: This study stopped at phase I and did not move forward to the phase II part.
Groups:
- Phase II: This study stopped at phase I and did not move forward to the phase II part.
Arm/Group | Phase II
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Time Frame: Assessed every 3 months for 2 years
Population: This study stopped at phase I and did not move forward to the phase II part.
Arm/Group | Phase II
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Rate
Time Frame: Assessed every 3 months for 2 years
Population: This study stopped at phase I and did not move forward to the phase II part.
Arm/Group | Phase II
Number analyzed (Participants) | 0

6. Secondary Outcome: Disease Control Rate
Time Frame: Assessed every 3 months for 2 years
Population: This study stopped at phase I and did not move forward to the phase II part.
Arm/Group | Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Description: All patients are included in the analyses of all-cause mortality and adverse events.
Groups:
- Arm A (Phase I - Initial Dose Level): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Patients also receive WEE1 inhibitor MK-1775 PO daily on days 1, 2, 8, 9, 15, and 16.
- Arm B (Phase I - Dose Level -2): Patients receive paclitaxel albumin-stabilized nanoparticle formulation, gemcitabine hydrochloride, and WEE1 inhibitor MK-1775 as in Arm A.
Arm/Group | Arm A (Phase I - Initial Dose Level) | Arm B (Phase I - Dose Level -2)
All-Cause Mortality (participants affected / at risk) | 2/2 | 5/5
Serious Adverse Events (participants affected / at risk) | 2/2 | 5/5
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Phase I - Initial Dose Level) (N=2) | Arm B (Phase I - Dose Level -2) (N=5)
Anemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Phase I - Initial Dose Level) (N=2) | Arm B (Phase I - Dose Level -2) (N=5)
Anemia (Blood and lymphatic system disorders) | 2 | 3
Atrial fibrillation (Cardiac disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 5
Fever (General disorders) | 1 | 2
Pain (General disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 1 | 4
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3
Alkaline phosphatase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 2
Creatinine increased (Investigations) | 0 | 1
INR increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 3
Weight loss (Investigations) | 1 | 2
White blood cell decreased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Weight gain (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT02194829/Prot_SAP_000.pdf